CLINICAL TRIAL: NCT01743066
Title: Vitamin E Level in Buccal Cells of Arsenicosis Patients Following Vitamin E Supplementation
Brief Title: Vitamin E Level in Buccal Cells of Arsenicosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Prof. Mir Misbahuddin, Prof. and Chairman, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BSMMU-004-CT
Record Dates: First submitted 2012-12-01; First posted 2012-12-06 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Chronic Arsenic Poisoning
Keywords: Arsenic; Arsenicosis; Buccal cells; Serum; Vitamin E; Cholesterol
MeSH Terms: interventions — Vitamin E

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arsenicosis patients (Experimental): Vitamin E (200 IU, caplet) daily orally for 20 weeks
  Interventions: Dietary Supplement: Vitamin E
- Arsenic exposed controls (Active Comparator): vitamin E (200 IU, caplet) daily orally for 20 weeks
  Interventions: Dietary Supplement: Vitamin E
- Heathy volunteers (Active Comparator): Vitamin E (200 IU, caplet) daily orally for 20 weeks
  Interventions: Dietary Supplement: Vitamin E

INTERVENTIONS:
Dietary Supplement: Vitamin E — vitamin E (200 IU, caplet) daily orally for 20 weeks

SUMMARY:
To understand the pathogenesis of chronic arsenic toxicity, the investigators need to know the levels of vitamin E in patients chronically exposed to high concentration of arsenic and if changes are found, what happens when supplemented with vitamin E. The buccal cells and serum of patients will be collected for the estimation of vitamin E both before and after supplementation with vitamin E. Similar samples will be collected from similar number of arsenic exposed controls and healthy volunteers for comparison.

DETAILED DESCRIPTION:
Chronic consumption of arsenic through water (drinking and cooking) and food leads to accumulation of arsenic within the cell. We usually give emphasis on the skin manifestations (melanosis and keratosis) of arsenicosis that is diagnosed first. Other manifestations remain un-diagnosed or diagnosed later. The severe form is the development of cancer in different organs mainly skin, lungs and urinary bladder. To understand the pathophysiology of the development of clinical manifestations appearing in the skin first, we need to understand interior of cells other than skin. One of the dietary supplements, vitamin E is found to be effective in improving the clinical signs/symptoms of melanosis and keratosis. Buccal cells are also exposed to arsenic and easy to collect. To understand the pathogenesis, we need to know the levels of vitamin E in patients of arsenicosis and if changes, what happens when supplemented with vitamin E. The buccal cells and serum of 20 patients will be collected for the estimation of vitamin E both before and after supplementation with vitamin E (200 IU, caplet) daily orally for 20 weeks. Similar samples will be collected from 20 arsenic exposed controls and 20 healthy volunteers for comparison.

ELIGIBILITY:
Inclusion Criteria:

For arsenicosis

* who drank arsenic contaminated water (>50 µg/L) for more than 6 months
* having physical signs of moderate degree of melanosis and keratosis

For arsenic exposed control

* relative or family member of the patient
* showing no physical signs of melanosis and keratosis
* share same tube well water for drinking purpose for more than 6 months

For healthy volunteers

* who drank arsenic safe water (<50 µg/L)
* live in the same Upazilla
* have no cutaneous manifestation
* who voluntarily agree to participate

Exclusion Criteria:

* tuberculosis, eczema psoriasis, contact dermatitis
* patients getting treatment of arsenicosis
* subject who voluntarily do not agree to participate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change in the amount of vitamin E in buccal cells | 0 week (baseline), 20 weeks (end)
  Changes in the amount of vitamin E in buccal cells of arsenicosis patients, arsenic exposed controls and healthy volunteers will be estimated both before and after supplementation with vitamin E for 20 weeks.

SECONDARY OUTCOMES:
Changes in the amount of cholesterol in buccal cells | 0 week (baseline), 20 weeks (end)
  Changes in the amount of cholesterol in buccal cells of arsenicosis patients, arsenic exposed controls and healthy volunteers will be estimated both before and after supplementation with vitamin E for 20 weeks.
Changes in the concentration of vitamin E in serum | 0 week (baseline), 20 weeks (end)
  Changes in the concentration of vitamin E in serum of arsenicosis patients, arsenic exposed controls and healthy volunteers will be estimated both before and after supplementation with vitamin E for 20 weeks.
Changes in the concentration of cholesterol in serum | 0 week (baseline), 20 weeks (end)
  Changes in the concentration of cholesterol in serum of arsenicosis patients, arsenic exposed controls and healthy volunteers will be estimated both before and after supplementation with vitamin E for 20 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pharmacology, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh